CLINICAL TRIAL: NCT02772783
Title: Dietary Glycemic Index, Brain Function and Food Intake in Patients With Type 1 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Belinda Lennerz, Instructor in Pediatric Endocrinology, Boston Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-P00022176; IRB- 2016P000079 (Other: Beth Israel Deaconess Medical Center)
Record Dates: First submitted 2016-05-11; First posted 2016-05-16 (Estimated); Results first posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-05

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: brain; fMRI; carbohydrate; insulin clamp; intake regulation; overweight; glycemic index
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Overweight

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- high GI meal, euglycemic insulin clamp (Experimental): A nutritional shake with high GI will be consumed. Regular insulin will be administered intravenously according to a negative feedback algorithm to maintain euglycemia.This condition results in euglycemia with high insulin levels.
  Interventions: Other: high GI meal; Drug: euglycemic insulin clamp
- high GI meal, fixed insulin infusion (Experimental): A nutritional shake with high GI will be consumed. Regular insulin will be administered intravenously at a rate previously established to maintain euglycemia after a low glycemic index meal. This condition results in moderate hyperglycemia with low insulin levels.
  Interventions: Other: high GI meal; Drug: primed-variable insulin infusion
- low GI meal, euglycemic insulin clamp (Active Comparator): A nutritional shake with low GI will be consumed. Regular insulin will be administered intravenously according to a negative feedback algorithm to maintain euglycemia. This condition results in euglycemia with low insulin levels.
  Interventions: Other: low GI meal; Drug: euglycemic insulin clamp

INTERVENTIONS:
Other: high GI meal — High and low GI liquid test meals are matched for macronutrient composition (60% carbohydrate, 15% protein, 25% fat), micronutrient profiles, physical properties, palatability and sweetness. Meals will provide 25% of individual daily energy requirements as estimated by the Harris Benedict equation. A high glycemic index of ~90 is achieved by using corn syrup as a carbohydrate source.
  Arms: high GI meal, euglycemic insulin clamp; high GI meal, fixed insulin infusion
Other: low GI meal — High and low GI liquid test meals are matched for macronutrient composition (60% carbohydrate, 15% protein, 25% fat), micronutrient profiles, physical properties, palatability and sweetness. Meals will provide 25% of individual daily energy requirements as estimated by the Harris Benedict equation. A low glycemic index of ~40 is achieved by using uncooked corn starch as a carbohydrate source.
  Arms: low GI meal, euglycemic insulin clamp
Drug: euglycemic insulin clamp — Insulin will be given intravenously for 5 hours. During the entire clamp protocol, glucose levels will be measured every 5 minutes. A basal insulin infusion will be started at 80% of the patients insulin pump basal rate, and will be adjusted between 0.1 and 2.5 mU/kg•min, depending upon the patient's plasma glucose level in relation to the target range target of 90-100 mg/dl.
  Arms: high GI meal, euglycemic insulin clamp; low GI meal, euglycemic insulin clamp
Drug: primed-variable insulin infusion — A primed-variable infusion of insulin will be administered at the rate established to achieve euglycemia after a low glycemic index meal. This is expected to result in moderate hyperglycemia as the high GI meal is associated with higher insulin requirements. For patient safety, glucose levels will be measured every 30 minutes. If glucose levels are > 400 mg/dl or < 60 mg/dl, insulin infusion will be adjusted to maintain glucose levels target of 60-400 mg/dl.
  Arms: high GI meal, fixed insulin infusion

SUMMARY:
Processed carbohydrates cause rapid changes in blood sugar and have been associated with overeating and obesity. We have shown that test meals high in processed carbohydrate affect brain areas involved in addiction, craving and overeating. It is unknown whether the changes in blood sugar or the associated higher insulin levels mediate this brain activation and its likely adverse effects.

Answering this question is important for patients with type 1 diabetes who have elevated risks of obesity and disordered eating: If blood sugar is the causal mechanism, optimal insulin coverage should be protective. If insulin is the causal mechanism, however, a diet high in processed carbohydrate could predispose to overeating and weight gain, as this diet requires higher insulin doses.

To disentangle these factors, we will study brain activation and relevant blood markers in 15 men with diabetes. In 4 sessions, we will examine meals with differential carbohydrate properties while giving insulin infusions.

DETAILED DESCRIPTION:
A total of 15 male participants (age 18-45) with T1DM will be recruited. Participants will be enrolled in the study for a total of 1-3 months, and participate in a pre-test visit and three test visits, each after a 10-12-hr overnight fast. Participants will be instructed to consume their regular, weight maintaining diet between visits.

At the pre-test visit, the study director or PI will meet participants, confirm eligibility and obtain informed consent. Participants will receive a low glycemic index (GI) meal with optimal iv insulin coverage using a negative feedback algorithm to maintain euglycemia (euglycemic clamp). Insulin requirement will be quantified. At some time during the visit, participants will present to the BIDMC research imaging facility for a practice MRI session, during which they will undergo a brief imaging sequence to get accustomed to the scanning process and eliminate anxiety as a confounder of imaging data.

At each of 3 test visits, one of the following experimental conditions will be applied in a randomized, blinded cross-over design: (a) high GI meal with euglycemic clamp, (b) low GI meal with euglycemic clamp, (c) high GI meal with primed-variable insulin infusion at the rate established during the pre-test visit. After steady state is established, baseline laboratory evaluation and MRI imaging will be obtained, followed by the test meal. Imaging will be repeated at 1 and 4 hours postprandial. Blood samples for pertinent metabolic and hormonal parameters will be obtained every 30 minutes. Each test-visit concludes with a standard weighed meal to quantify ad-libitum intake.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for a minimum of 3 years
* BMI 20-35 kg/m2
* Use of insulin pump
* Willing and able to: Maintain weight and document for duration of the study

Exclusion Criteria:

* Insulin resistance (current insulin requirement > 1.5 U/kg/d)
* Insulin requirement < 0.5 unit/kg/day (cut-off for preserved beta-cell function)
* HbA1C ≥ 8.0%
* DKA within 2 months
* Frequent hypoglycemia (BG <50 mg/dl), > 3 times per week
* Fluctuations in body weight >10% over preceding year
* Smoking or illicit substance abuse
* High levels of physical activity (≥60 minutes per day, ≥ 4 days per week)
* Current weight loss diet
* Medical problems, medications or dietary supplements that may affect metabolism, insulin action, body weight, appetite, energy expenditure, or gastrointestinal absorption (e.g. celiac disease)
* Allergies to compounds or intolerance of the liquid meals
* MRI exclusion criteria
* Other conditions according to self-report that would prohibit participation based and researcher assessment

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2016-07; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Belinda S Lennerz, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Boston Children's Hospital Diabetes Program and via postings in the surrounding medical area.
Pre-assignment Details: Participants underwent a 5 hour pre-randomization visit to establish IV insulin requirement for a low GI test meal. Participants were positioned in the MRI scanner for a brief test sequence.
  Participants were excluded if they were unable to finish these pre-randomization procedures, or if they decided to not continue.
Groups:
- High GI Matched Glucose - Low GI - High GI Matched Insulin: In a randomized cross-over design, a nutritional shake with high GI vs low GI was consumed with differential insulin coverage in the following order:
  1. High GI meal covered with IV insulin adjusted using a negative feedback algorithm to achieve euglycemia, resulting in hyperinsulinemia (experimental condition A); 1 day.
     - 1-week wash-out
  2. Low GI meal covered with IV insulin adjusted using a negative feedback algorithm to achieve euglycemia (comparison condition B); 1 day.
     - 1-week wash-out
  3. High GI meal with IV insulin matching the low GI meal, resulting in hyperglycemia (experimental condition C); 1 day.
  High and low GI liquid test meals were matched for macronutrient composition (60% carbohydrate, 15% protein, 25% fat), micronutrient profiles, physical properties, palatability and sweetness. Meals provided 25% of individual daily energy requirements.
  Insulin was given intravenously for 5 hours. Glucose levels were measured every 5 minutes for insulin titration.
- High GI Matched Insulin - Low GI - High GI Matched Glucose: In a randomized cross-over design, a nutritional shake with high GI vs low GI was consumed with differential insulin coverage in the following order:
  1. High GI meal with IV insulin matching the low GI meal (as determined during the pre-randomization visit), resulting in hyperglycemia (experimental condition C); 1 day.
     - 1-week wash-out
  2. Low GI meal covered with IV insulin adjusted using a negative feedback algorithm to achieve euglycemia (comparison condition B); 1 day.
     - 1-week wash-out
  3. High GI meal covered with IV insulin adjusted using a negative feedback algorithm to achieve euglycemia, resulting in hyperinsulinemia (experimental condition A); 1 day.
  High and low GI liquid test meals were matched for macronutrient composition (60% carbohydrate, 15% protein, 25% fat), micronutrient profiles, physical properties, palatability and sweetness. Meals provided 25% of individual daily energy requirements.
  Insulin was given intravenously for 5 hours. Glucose levels were measured every 5 minutes for insulin titration.
Period: Experimental Condition 1, 1 Day
Arm/Group | High GI Matched Glucose - Low GI - High GI Matched Insulin | High GI Matched Insulin - Low GI - High GI Matched Glucose
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0
Period: Wash-out, 1 Week
Arm/Group | High GI Matched Glucose - Low GI - High GI Matched Insulin | High GI Matched Insulin - Low GI - High GI Matched Glucose
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0
Period: Comparison Condition, 1 Day
Arm/Group | High GI Matched Glucose - Low GI - High GI Matched Insulin | High GI Matched Insulin - Low GI - High GI Matched Glucose
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0
Period: Wash-out, 1 Week
Arm/Group | High GI Matched Glucose - Low GI - High GI Matched Insulin | High GI Matched Insulin - Low GI - High GI Matched Glucose
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0
Period: Experimental Condition 2, 1 Day
Arm/Group | High GI Matched Glucose - Low GI - High GI Matched Insulin | High GI Matched Insulin - Low GI - High GI Matched Glucose
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: In a randomized cross-over design, a nutritional shake with high GI vs low GI was consumed with differential insulin coverage:
  * High GI meal covered with IV insulin to to achieve euglycemia, resulting in hyperinsulinemia (experimental condition A); 1 day.
  * 1-week wash-out
  * Low GI meal covered with IV insulin to achieve euglycemia (comparison condition B); 1 day.
  * 1-week wash-out
  * High GI meal with IV insulin matching the low GI meal, resulting in hyperglycemia (experimental condition A); 1 day.
  The order of experimental conditions A and B was randomized.
  High and low GI liquid test meals were matched for macronutrient composition (60% carbohydrate, 15% protein, 25% fat), micronutrient profiles, physical properties, palatability and sweetness. Meals provided 25% of individual daily energy requirements.
  Insulin was given intravenously for 5 hours. Glucose levels were measured every 5 minutes for insulin titration.
  Because all participants completed all interventions, results are presented in aggregate for the entire study group.
Arm/Group | All Study Participants
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 21 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15
BMI [Mean (Standard Deviation); unit: kg/m^2] | 21 (1.4)

OUTCOME MEASURES:

1. Primary Outcome: Nucleus Accumbens Blood Flow
Description: Cerebral blood flow in the right and left nucleus accumbent was measured by arterial spin labeling (MRI). Blood flow was normalized for whole brain perfusion and corrected for baseline perfusion in the respective brain area and meal order, as per our a priori statistical analysis plan.
Time Frame: 4 hrs postprandial
Measure: Least Squares Mean (Standard Error); unit: ml/g/min per ml/g/min
Groups:
- High GI With Matched to Low GI Glucose (HGI HI): After an overnight fast, a nutritional shake with high GI was consumed. The shake provided 25% of daily calorie requirements with a macronutrient composition of 60% carbohydrate, 15% protein, 25% fat, and matched micronutrient profiles, physical properties, palatability and sweetness.
  Insulin was given intravenously to normalize blood glucose before the meal and for 5 hours postprandial. Blood glucose levels were measured every 5 minutes, and Insulin was adjusted using a negative feedback algorithm to maintain euglycemia.
  Interventions were presented in a cross-over design. Because all participants completed all interventions, results are presented by intervention.
- Low GI (LGI): After an overnight fast, a nutritional shake with low GI was consumed. The shake provided 25% of daily calorie requirements with a macronutrient composition of 60% carbohydrate, 15% protein, 25% fat, and matched micronutrient profiles, physical properties, palatability and sweetness.
  Insulin was given intravenously to normalize blood glucose before the meal and for 5 hours postprandial. Blood glucose levels were measured every 5 minutes, and Insulin was adjusted using a negative feedback algorithm to maintain euglycemia.
  Interventions were presented in a cross-over design. Because all participants completed all interventions, results are presented by intervention.
- High GI With Matched to Low GI Insulin (HGI LI): After an overnight fast, a nutritional shake with high GI was consumed. The shake provided 25% of daily calorie requirements with a macronutrient composition of 60% carbohydrate, 15% protein, 25% fat, and matched micronutrient profiles, physical properties, palatability and sweetness.
  Insulin was given intravenously to normalize blood glucose before the meal and for 5 hours postprandial. Blood glucose levels were measured every 5 minutes. Insulin was given at the same rates as determined appropriate for each participant during the pre-randomization visit or the LGI visit.
  Interventions were presented in a cross-over design. Because all participants completed all interventions, results are presented by intervention.
Arm/Group | High GI With Matched to Low GI Glucose (HGI HI) | Low GI (LGI) | High GI With Matched to Low GI Insulin (HGI LI)
Number analyzed (Participants) | 15 | 15 | 15
ml/g/min per ml/g/min
  right | 1.13 (0.02) | 1.16 (0.02) | 1.15 (0.02)
  left | 1.21 (0.02) | 1.18 (0.02) | 1.18 (0.02)

2. Secondary Outcome: Nucleus Accumbens Blood Flow
Description: as for outcome 1
Time Frame: 1 hr postprandial
Measure: Least Squares Mean (Standard Error); unit: ml/g/min per ml/g/min
Arm/Group | High GI With Matched to Low GI Glucose (HGI HI) | Low GI (LGI) | High GI With Matched to Low GI Insulin (HGI LI)
Number analyzed (Participants) | 15 | 15 | 15
ml/g/min per ml/g/min
  right | 1.12 (0.02) | 1.16 (0.02) | 1.11 (0.02)
  left | 1.20 (0.02) | 1.19 (0.02) | 1.14 (0.02)

3. Secondary Outcome: Blood Flow in Other Brain Areas Involved in Intake Regulation - Dorsal Caudate
Description: Cerebral blood flow was measured by arterial spin labeling (MRI). Grouped MRI data was visually inspected for postprandial differences between conditions. Blood flow from a cluster contracting the conditions in the right dorsal caudate, just lateral to the nucleus accumbent, was extracted, normalized for whole brain perfusion and corrected for baseline perfusion in the respective brain area and meal order, as per our a priori statistical analysis plan.
Time Frame: 4 hrs postprandial
Measure: Least Squares Mean (Standard Error); unit: ml/g/min per ml/g/min
Arm/Group | High GI With Matched to Low GI Glucose (HGI HI) | Low GI (LGI) | High GI With Matched to Low GI Insulin (HGI LI)
Number analyzed (Participants) | 15 | 15 | 15
ml/g/min per ml/g/min | 0.60 (0.01) | 0.59 (0.01) | 0.64 (0.01)

4. Secondary Outcome: Blood Flow in Other Brain Areas Involved in Intake Regulation - Ventrolateral Striatum
Description: Cerebral blood flow was measured by arterial spin labeling (MRI). Grouped MRI data was visually inspected for postprandial differences between conditions. Blood flow from a cluster contracting the conditions in the right ventrolateral striatum, just lateral to the nucleus accumbent, was extracted, normalized for whole brain perfusion and corrected for baseline perfusion in the respective brain area and meal order, as per our a priori statistical analysis plan.
Time Frame: 1 hr postprandial
Measure: Least Squares Mean (Standard Error); unit: ml/g/min per ml/g/min
Arm/Group | High GI With Matched to Low GI Glucose (HGI HI) | Low GI (LGI) | High GI With Matched to Low GI Insulin (HGI LI)
Number analyzed (Participants) | 15 | 15 | 15
ml/g/min per ml/g/min | 0.60 (0.01) | 0.61 (0.01) | 0.60 (0.01)

5. Secondary Outcome: Functional Connectivity of Nucleus Accumbens, Hypothalamus and Other Brain Areas Involved in Intake Regulation
Description: Cerebral blood oxygen concentration level was measured by resting state functional MRI (rs-fMRI). Seed based analysis was performed with the seed on the right Nucleus Accumbens. Functional connectivity between Nucleus Accumbens and Hypothalamus was assessed through extraction of temporal correlation measures.
Time Frame: 4 hrs postprandial
Measure: Least Squares Mean (Standard Error); unit: unite-less correlation
Arm/Group | High GI With Matched to Low GI Glucose (HGI HI) | Low GI (LGI) | High GI With Matched to Low GI Insulin (HGI LI)
Number analyzed (Participants) | 13 | 13 | 13
unite-less correlation | 0.26 (0.08) | 0.24 (0.08) | 0.25 (0.08)

6. Secondary Outcome: Functional Connectivity of Nucleus Accumbens, Hypothalamus and Other Brain Areas Involved in Intake Regulation
Description: Cerebral blood oxygen concentration level was measured by resting state functional MRI (rs-fMRI). Seed based analysis was performed with the seed on the right Nucleus Accumbens. Functional connectivity between Nucleus Accumbens and Hypothalamus was assessed through extraction of temporal correlation measures. Functional connectivity between Nucleus Accumbens and other brain areas was visually assessed.
Time Frame: 1 hr postprandial
Measure: Least Squares Mean (Standard Error); unit: unite-less correlation
Arm/Group | High GI With Matched to Low GI Glucose (HGI HI) | Low GI (LGI) | High GI With Matched to Low GI Insulin (HGI LI)
Number analyzed (Participants) | 13 | 13 | 13
unite-less correlation | 0.36 (0.09) | 0.15 (0.09) | 0.15 (0.09)

7. Other Pre Specified Outcome: Plasma Glucose Level
Description: blood samples will be obtained every 30 minutes
Time Frame: 0-4.5 hrs postprandial
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Serum Insulin Level
Description: blood samples will be obtained every 30 minutes
Time Frame: 0-4.5 hrs postprandial
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Serum Fatty Acids
Description: blood samples will be obtained every 30 minutes
Time Frame: 0-4.5 hrs postprandial
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Plasma Ghrelin
Description: blood samples will be obtained every 30 minutes and analyzed as part of a metabolic hormone panel
Time Frame: 0-4.5 hrs postprandial
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Plasma GLP-1
Description: blood samples will be obtained every 30 minutes and analyzed as part of a metabolic hormone panel
Time Frame: 0-4.5 hrs postprandial
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Plasma PYY
Description: blood samples will be obtained every 30 minutes and analyzed as part of a metabolic hormone panel
Time Frame: 0-4.5 hrs postprandial
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Plasma CCK
Description: analyzed as part of a metabolic hormone panel
Time Frame: 0-4.5 hrs postprandial
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Plasma Glucagon
Description: blood samples will be obtained every 30 minutes and analyzed as part of a metabolic hormone panel
Time Frame: 0-4.5 hrs postprandial
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Plasma Leptin
Description: analyzed as part of a metabolic hormone panel
Time Frame: 0-4.5 hrs postprandial
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Metabolomics
Description: LC-MS/MS methodology using several chromatographic stationary phases for > 400 metabolites
Time Frame: 0, 1 and 4 hrs postprandial
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Enrollment through study completion (on average 2 months).
Groups:
- High GI With Matched to Low GI Glucose (HGI HI): After an overnight fast, a nutritional shake with high GI was consumed. The shake provided 25% of daily calorie requirements with a macronutrient composition of 60% carbohydrate, 15% protein, 25% fat, and matched micronutrient profiles, physical properties, palatability and sweetness.
  Insulin was given intravenously to normalize blood glucose before the meal and for 5 hours postprandial. Blood glucose levels were measured every 5 minutes, and Insulin was adjusted using a negative feedback algorithm to maintain euglycemia.
- Low GI (LGI): After an overnight fast, a nutritional shake with low GI was consumed. The shake provided 25% of daily calorie requirements with a macronutrient composition of 60% carbohydrate, 15% protein, 25% fat, and matched micronutrient profiles, physical properties, palatability and sweetness.
  Insulin was given intravenously to normalize blood glucose before the meal and for 5 hours postprandial. Blood glucose levels were measured every 5 minutes, and Insulin was adjusted using a negative feedback algorithm to maintain euglycemia.
- High GI With Matched to Low GI Insulin (HGI LI): After an overnight fast, a nutritional shake with high GI was consumed. The shake provided 25% of daily calorie requirements with a macronutrient composition of 60% carbohydrate, 15% protein, 25% fat, and matched micronutrient profiles, physical properties, palatability and sweetness.
  Insulin was given intravenously to normalize blood glucose before the meal and for 5 hours postprandial. Blood glucose levels were measured every 5 minutes. Insulin was given at the same rates as determined appropriate for each participant during the pre-randomization visit or the LGI visit.
Arm/Group | High GI With Matched to Low GI Glucose (HGI HI) | Low GI (LGI) | High GI With Matched to Low GI Insulin (HGI LI)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 1/15 | 0/15 | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High GI With Matched to Low GI Glucose (HGI HI) (N=15) | Low GI (LGI) (N=15) | High GI With Matched to Low GI Insulin (HGI LI) (N=15)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
dizzyness (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-26): https://cdn.clinicaltrials.gov/large-docs/83/NCT02772783/Prot_SAP_000.pdf